CLINICAL TRIAL: NCT01197885
Title: International, Multicenter, Open-label, Phase II Study to Investigate the Efficacy and Safety of Multiple Doses of IMAB362 in Patients With Advanced Adenocarcinoma of the Stomach or the Lower Esophagus
Brief Title: Efficacy and Safety Study of Multiple Doses of IMAB362 in Patients With Advanced Gastroesophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ganymed Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GM-IMAB-001-02; 2009-017365-36 (EudraCT Number)
Record Dates: First submitted 2010-09-06; First posted 2010-09-09 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors
MeSH Terms: interventions — zolbetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMAB362 (Experimental): Two different doses (antibody / body surface area) of IMAB362 will be administered sequentially.
  Interventions: Drug: IMAB362

INTERVENTIONS:
Drug: IMAB362 — Cohort 1 repeated doses of 300 mg/m2 Cohort 2 repeated doses of 600 mg/m2 Cohort 3 doses to be determined, 600mg/m2 or less

SUMMARY:
IMAB362 is a monoclonal antibody specific for gastric or lower esophageal adenocarcinoma. Preclinically IMAB362 was shown to inhibit tumor growth and to kill cancer cells by indirect (complement-dependent cytotoxicity, antibody-dependent cellular cytotoxicity) and direct mechanisms (antiproliferative and proapoptotic effects). The aim of this phase II study is to establish efficacy and safety of multiple doses of IMAB362 as monotherapy in patients suffering from metastatic, refractory or recurrent adenocarcinoma of the stomach or the lower esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, refractory or recurrent disease of advanced adenocarcinoma of the stomach or the lower esophagus proven by histology
* CLDN18.2 expression of the biopsy material from the cancer confirmed by immunohistochemistry
* At least 1 measurable site of disease according to RECIST criteria

Exclusion Criteria:

* Less than 3 weeks since prior chemo-or radiation therapy
* Other concurrent anticancer therapies
* Concurrent anticoagulation with vitamin K antagonists
* Therapeutic doses of Heparin (prophylactic doses accepted)
* Uncontrolled or severe illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-09-03 (Actual); Primary Completion 2015-08-13 (Actual); Study Completion 2015-08-13 (Actual)

PRIMARY OUTCOMES:
Rate of remission (CR, PR) according to RECIST Criteria | All patients will be evaluated in 8-12 weeks intervals until 6 months after last infusion

SECONDARY OUTCOMES:
Number of Participants with adverse events as a measure of safety and tolerability | All patients will be evaluated in 8-12 weeks intervals until 6 months after last infusion
Frequency and severity of adverse events according to CTCAE v3.0 | All patients will be evaluated in 8-12 weeks intervals until 6 months after last infusion
Progression-free-survival time (PFS) | All patients will be evaluated in 8-12 weeks intervals until 6 months after last infusion
  The time from start of the first infusion to date of first observed disease progression or death due to progression (whichever is first)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schuler, Prof. Dr. med., Principal Investigator — Innere Klinik Universitätsklinikum Essen
Locations (21):
- Bulgaria (3):
  - Oncology Dispensary "Dr. Marko Markov", Varna
  - MHAT "St.Marina", Varna
  - Complex Oncology Center, Veliko Tarnovo
- Germany (13):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Medizinische Univeritätsklinik Ruhr-Universität Bochum, Bochum
  - Klinikum Braunschweig, Braunschweig
  - Universitätsklinikum Essen, Innere Klinik (Tumorforschung), Essen
  - Krankenhaus Nordwest, Klinik für Onkologie und Hämatologie, Frankfurt
  - Universitätsklinikum Halle, Halle
  - Universitäres Cancer Center Universitätsklinikum Eppendorf, Hamburg
  - Onkologische Schwerpunktpraxis Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, NCT, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin der Johannes-Gutenberg Universität, Mainz
  - Klinikum rechts der Isar, München
  - Universitätsklinikum Ulm, Ulm
- Latvia (3):
  - Piejuras Hospital, Liepāja
  - Paula Stradina Clinical University Hospital, Riga
  - Riga East Clinical Research, Riga
- Vilnius University, Vilnius, Lithuania
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Tureci O, Sahin U, Schulze-Bergkamen H, Zvirbule Z, Lordick F, Koeberle D, Thuss-Patience P, Ettrich T, Arnold D, Bassermann F, Al-Batran SE, Wiechen K, Dhaene K, Maurus D, Gold M, Huber C, Krivoshik A, Arozullah A, Park JW, Schuler M. A multicentre, phase IIa study of zolbetuximab as a single agent in patients with recurrent or refractory advanced adenocarcinoma of the stomach or lower oesophagus: the MONO study. Ann Oncol. 2019 Sep 1;30(9):1487-1495. doi: 10.1093/annonc/mdz199. PMID 31240302
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/GM-IMAB-001-02/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25769&tenant=MT_AST_9011
- See also: Updated Vivli Worksheet — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217491&parentIdentifier=GM-IMAB-001-02&attachmentIdentifier=0006468b-c70f-4556-b505-d281ac1aaa06&fileName=GM-IMAB-001-02_Data_Sharing_Platform_(Vivli)_Worksheet_16_Dec_2024.docx&versionIdentifier=